CLINICAL TRIAL: NCT05615012
Title: An Open-Label, Single-Sequence Crossover, Drug-Drug Interaction Study to Assess the Effect of Steady-State BMS-986322 on the Pharmacokinetics of Rosuvastatin (Part 1), the Pharmacokinetics and Pharmacodynamics of Metformin (Part 2) and the Pharmacokinetics of Methotrexate (Part 3) in Healthy Participants
Brief Title: A Study Investigating Interactions Between BMS-986322 and Rosuvastatin, Metformin and Methotrexate in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM032-039
Record Dates: First submitted 2022-11-07; First posted 2022-11-14 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Healthy Participants
Keywords: BMS-986322; Rosuvastatin; Metformin; Methotrexate
MeSH Terms: interventions — Rosuvastatin Calcium; Metformin; Glucose; Methotrexate; Leucovorin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1: Rosuvastatin + BMS-986322 (Experimental)
  Interventions: Drug: BMS-986322; Drug: Rosuvastatin
- Part 2: Metformin + BMS-986322 + Glucose (Experimental)
  Interventions: Drug: BMS-986322; Drug: Metformin; Dietary Supplement: Glucose
- Part 3: Methotrexate + BMS-986322 + Leucovorin (Experimental)
  Interventions: Drug: BMS-986322; Drug: Methotrexate; Drug: Leucovorin

INTERVENTIONS:
Drug: BMS-986322 — Specified dose on specified days
Drug: Rosuvastatin — Specified dose on specified days
  Arms: Part 1: Rosuvastatin + BMS-986322
Drug: Metformin — Specified dose on specified days
  Arms: Part 2: Metformin + BMS-986322 + Glucose
Dietary Supplement: Glucose — Specified dose on specified days
  Arms: Part 2: Metformin + BMS-986322 + Glucose
Drug: Methotrexate — Specified dose on specified days
  Arms: Part 3: Methotrexate + BMS-986322 + Leucovorin
Drug: Leucovorin — Specified dose on specified days
  Arms: Part 3: Methotrexate + BMS-986322 + Leucovorin

SUMMARY:
The aim of this study is to assess the effect of coadministration of multiple oral doses of BMS-986322 with rosuvastatin, metformin, and methotrexate in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator, a healthy participant, as determined by no clinically significant deviation from normal in medical history, physical examination, ECGs, and clinical laboratory determinations.
* Body mass index (BMI) of 18.0 kilogram (kg)/meter(m)^2 to 30.0 kg/m^2, inclusive, and body weight ≥ 50 kg for males and ≥ 45 kg for females, at screening.
* A female participant is eligible to participate if she is a woman not of childbearing potential.
* Female participants must refrain from donating oocytes during the intervention period and for at least 5 half-lives (5 days) after the last dose of study intervention.
* For Parts 1 and 2 participants must be 18 to 60 years of age.
* For Part 3 participants must be 18 to 50 years of age.

Exclusion Criteria:

* Any significant acute or chronic medical illness.
* Any major surgery, including any gastrointestinal (GI) surgery, with the exception of appendectomy, within 90 days of study intervention administration.
* History of alcohol abuse within 1 year prior to screening or regular use of alcohol within 6 months prior to screening that exceeds 7 units for women or 14 units for men of alcohol per week (1 unit = 340 mililitre [mL] of beer 5%, 140 mL of wine 12%, or 45 mL of distilled alcohol 40%).
* Participant must not have a known or suspected immune-mediated disorder, or any history of known or suspected congenital or acquired immunodeficiency state or condition that would compromise the participant's immune status.
* Participant must not have any history or risk for tuberculosis (TB) in participants with current clinical, radiographic, or laboratory evidence of active TB.

Other protocol-defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 21 days
Area under the plasma concentration-time curve from time zero extrapolated to infinite time (AUC[INF]) | Up to 21 days
Area under the plasma concentration-time curve from time zero to time of last quantifiable concentration (AUC [0-T]) | Up to 21 days

SECONDARY OUTCOMES:
Time of maximum observed plasma concentration (Tmax) | Up to 21 days
Apparent terminal phase half-life (T-HALF) | Up to 21 days
Apparent total body clearance (CLT/F) | Up to 21 days
Number of participants with adverse events (AEs) | Up to 51 days
Number of participants with vital sign abnormalities | Up to 51 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 51 days
Number of participants with physical examination abnormalities | Up to 51 days
Number of participants with clinical laboratory abnormalities | Up to 51 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html